CLINICAL TRIAL: NCT05320601
Title: Efficacy of Peripheral Magnetic Stimulation Compare to Dry Needling in Patient With Upper Trapezius Myofascial Pain Syndrome
Brief Title: Efficacy of Peripheral Magnetic Stimulation Compare to Dry Needling in Myofascial Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Apiphan Iamchaimongkol, MD, Principal Investigator, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AIamchaimongkol
Record Dates: First submitted 2022-03-25; First posted 2022-04-11 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-07

CONDITIONS: Myofascial Pain Syndrome
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Repetitive Peripheral Magnetic Stimulation (Experimental): Repetitive Peripheral Magnetic Stimulation 1 session
  Interventions: Device: Repetitive Peripheral Magnetic Stimulation
- Dry Needling (Experimental): Dry Needling 1 session
  Interventions: Procedure: Dry needling

INTERVENTIONS:
Device: Repetitive Peripheral Magnetic Stimulation — Repetitive Peripheral Magnetic Stimulation at trigger point of upper trapezius muscle
  Arms: Repetitive Peripheral Magnetic Stimulation
Procedure: Dry needling — Dry needling at trigger point of upper trapezius muscle
  Arms: Dry Needling

SUMMARY:
Compare efficiency between repetitive peripheral magnetic stimulation and dry needling in patient with upper trapezius myofascial pain syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patients with myofascial pain syndrome at unilateral upper trapezius muscle and had pain score (Visual analog scale) at least 4

Exclusion Criteria:

* Patients with signs and/or symptoms of neurological deficit
* Patients with history of cervical hernia, cervical radiculopathy, cervical myelopathy, fibromyalgia, whiplash spondylosis and cervical spinal stenosis.
* Patients who received physical therapy/injection/surgery at neck or pain area in last 6 months.
* Patients with abnormal coagulopathy and/or currently use anticoagulant medicine.
* Patients with cardiac device.
* Patients with history of aneurysm clip procedure, stent-coils procedure or cochlear implant surgery.
* Pregnancy

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Change of Visual analog scale | Change from baseline Visual analog scale at immediately after intervention, Change from Baseline visual analog scale at 1 week and Change from baseline Visual analog scale at 4 weeks
  Pain measurement Score from 0-10, 0 means no pain and 10 means maximum pain. Higher scores mean worse outcome.

SECONDARY OUTCOMES:
Neck disability index | Change from baseline Neck disability index at immediately after intervention, Change from Baseline Neck disability index at 1 week and Change from baseline Neck disability index at 4 weeks
  Disability secondary to neck pain Score from 0-50, 0 means no disability and 50 means complete disability. Higher scores mean worse outcome.

OTHER OUTCOMES:
Pain pressure threshold | Change from baseline Pain pressure threshold at immediately after intervention, Change from Baseline Pain pressure threshold at 1 week and Change from baseline Pain pressure threshold at 4 weeks
  The minimum pressure that induces pain in trigger point. Higher scores mean better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Apiphan Iamchaimongkol, M.D., Study Director — Ramathibodi Hospital
Locations (1):
- Physical medicine and rehabilitation, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The effect of repetitive magnetic stimulation on localized musculoskeletal pain — https://pubmed.ncbi.nlm.nih.gov/9665594/